CLINICAL TRIAL: NCT01615094
Title: BNP and Neuroimmune Characteristics of CHF and Depression (Competing Renewal)
Brief Title: Cardiac Health, Mood, & Neuroimmune Activation
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Paul J. Mills, Professor IR, University of California, San Diego
Other Study IDs: 5R01HL073355-06 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure; Depression
MeSH Terms: conditions — Heart Failure; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High-risk Stage B Heart Failure Patients: American College of Cardiology/American Heart Association (ACC/AHA) asymptomatic Stage B patients with B-Type natriuretic peptide (BNP) ≥ 65pg/ml

SUMMARY:
The study is designed to find out more about how mood and the nervous system affect the body's immune system. The investigators plan to study this in people who have been identified by their physician as being at-risk for the development of heart failure. There will be approximately 525 individuals participating in this study at UCSD and at the VASDHS. Individuals who will be asked to take part in this study will have a functional or structural heart problem apparent on an echocardiogram, or a previous heart attack, but no symptoms of heart failure. Some individuals will only complete one assessment (consisting of psychological questionnaires and interview, walk test, blood draw, and body measurements), whereas others deemed "high-risk" on the basis of a laboratory test, will be asked to complete that same assessment every 6 months for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18 years or older
2. ACC/AHA classification Stage B HF patients
3. Receiving optimal treatment according to their cardiologist and/or internists
4. An echocardiogram within the past 12 months
5. Ejection fraction: as described below in Initial Screening and Identification of Stage B Patients
6. Men and women of all ethnicities and races
7. Ability and physician clearance to perform mild exercise
8. With and without depressive symptoms and DSM-IV MDD
9. Ability to fully understand all elements of and sign the written informed consent before initiation of the study

Exclusion Criteria:

1. History of recent myocardial infarction (3 months)
2. Significant aortic or mitral stenosis, angina not adequately managed with nitrates
3. Coronary revascularization, mitral valve repair or any other cardiac surgery or implantation of a biventricular pacemaker within the past 2 months
4. Hypertension >180/110 mm Hg
5. Recent stroke or significant cerebral neurological impairment
6. Severe COPD, patients who require mechanical ventilation, with cardiogenic shock, volume depletion
7. Subjects with high suicide risk
8. Immune-related disorders including infectious diseases and autoimmune and inflammatory disorders
9. Morbid Obesity: BMI > 40 due to likelihood of inability to perform exercise
10. Women who are pregnant or nursing
11. Major mental illness as determined by referring provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: American College of Cardiology/American Heart Association (ACC/AHA) asymptomatic Stage B patients with B-Type natriuretic peptide (BNP) ≥ 65pg/ml
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2011-01; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Rate of dysphoria | up to 4 years
  In high-risk (BNP ≥ 65pg/ml) Stage B patients, characterize rates of clinically significant depressed mood (BDI ≥10) and MDD (SCID) and determine prospective relationships with transition to Stages C and/or D HF and clinical outcomes during an average follow-up time of 30 months.

SECONDARY OUTCOMES:
Neuroimmune activation | up to 4 years
  In high-risk (BNP ≥ 65pg/ml) Stage B patients, characterize the role of neuroimmune activation (defined by circulating levels of C-reactive protein (CRP), Tumor Necrosis Factor-alpha (TNF-α), Interleukin (IL)-6, IL-1β, soluble intercellular adhesion molecule-1 (sICAM-1), soluble P-selectin (sP-selectin), norepinephrine, and functional leukocyte assays)in the relationship between clinically significant depressed mood and/or MDD and transition to symptomatic Stages C and/or D HF and clinical outcomes during an average follow-up time of 30 months.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Mills, PhD, Principal Investigator — University of California, San Diego

REFERENCES:
- [Derived] Redwine LS, Henry BL, Pung MA, Wilson K, Chinh K, Knight B, Jain S, Rutledge T, Greenberg B, Maisel A, Mills PJ. Pilot Randomized Study of a Gratitude Journaling Intervention on Heart Rate Variability and Inflammatory Biomarkers in Patients With Stage B Heart Failure. Psychosom Med. 2016 Jul-Aug;78(6):667-76. doi: 10.1097/PSY.0000000000000316. PMID 27187845